CLINICAL TRIAL: NCT04007120
Title: Open-label Study to Assess the Safety, Tolerability, Feasibility, and Pharmacokinetics of Inhaled RVT-1601 in Preterm Infants at High-risk for Long-term Respiratory Morbidities
Brief Title: Open-label Study of Inhaled RVT-1601 in Preterm Infants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Respivant Sciences GmbH (Industry)
Collaborators: Respivant Sciences Inc. (Industry)
Responsible Party: Sponsor
Organization: Respivant Sciences Inc. (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: RVT1601-RMP-01
Record Dates: First submitted 2019-06-28; First posted 2019-07-05 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Respiratory Morbidities of Prematurity (RMP)

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- RVT-1601 Low Dose (Experimental): Inhaled RVT-1601 administered once daily over two days via eFlow nebulizer
  Interventions: Drug: RVT-1601
- RVT-1601 Mid Dose (Experimental): Inhaled RVT-1601 administered once daily over two days via eFlow nebulizer
  Interventions: Drug: RVT-1601

INTERVENTIONS:
Drug: RVT-1601 — Inhaled RVT-1601 administered once daily over two days

SUMMARY:
Preterm birth predisposes infants to greater risk for respiratory morbidities and the need for pulmonary care compared to term infants both in the short-term and long-term. In the short-term, preterm birth is a high risk factor for development of bronchopulmonary dysplasia (BPD), the second most common chronic pediatric respiratory disease after asthma. In the long-term, following discharge from the neonatal intensive care unit (NICU) and the hospital, preterm birth carries a high risk for respiratory morbidities (e.g., wheezing, cough, doctor visits, and hospitalizations for respiratory infections) and resource use, which in turn predisposes infants to the development of lung diseases in childhood and adulthood, including airway hyperresponsiveness, asthma, and chronic obstructive pulmonary disease (COPD). There is a significant unmet need for safe and efficacious approaches in the prevention and treatment of respiratory morbidities of prematurity.

The study will be conducted in the neonatal intensive care unit (NICU) in preterm infants to determine safety, tolerability and lung delivery performance of RVT-1601, a new inhalation formulation of cromolyn sodium delivered via the eFlow® Closed System (CS) nebulizer/face mask.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants between 32 weeks 0 days and 34 weeks 6 days of PMA
* Born between 24 weeks 0 days and 29 weeks 6 days of estimated GA
* Requiring minimal or no respiratory support (i.e., supplemental oxygen with <2 liters per minute of nasal cannula flow acceptable)
* Body weight appropriate for gestational age
* Written informed consent obtained from at least one of the parents or legal guardians

Exclusion Criteria:

* Requiring invasive or noninvasive respiratory support (e.g., mechanical ventilation, CPAP)
* Clinically unstable (i.e. unable to maintain SpO2 between 90-95 % , escalating respiratory support in the past 24 hours)
* Major congenital anomaly (chromosomal, renal, cardiac, hepatic, neurologic or pulmonary malformations)
* Significant cardiac disorder (i.e., pulmonary hypertension)
* History of major surgical procedure
* Any condition that would preclude receiving study drug or performing any study-related procedures
* Participation in any other investigational drug study
* History of hypersensitivity or intolerance to cromolyn sodium

Ages: 32 Months to 35 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 8 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-05-29 (Actual); Study Completion 2020-05-29 (Actual)

PRIMARY OUTCOMES:
Change in heart rate | Pre-dose and 15 minutes post-dose
  Assessment of heart rate (beats/min)
Change in blood pressure | Pre-dose and 15 minutes post-dose
  Assessment of systolic and diastolic blood pressure (mmHg)
Change in oxygenation | Pre-dose and 15 minutes post-dose
  Assessment of peripheral capillary oxygen saturation (SpO2)

SECONDARY OUTCOMES:
Peak plasma concentration (Cmax) | 30 minutes post-dose
  Assessment of peak plasma concentration of RVT-1601
Total urine excretion | 8 hours post-dose
  Assessment of total urine content of RVT-1601

CONTACTS AND LOCATIONS:
Locations (1):
- Sharp Mary Birch Hospital for Women & Newborns, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No